CLINICAL TRIAL: NCT06832527
Title: Use of Virtual Reality to Improve Sensorimotor Function in Patients with Traumatic Wrist and Hand Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Leire Cruz-Gambero, Occupational therapist, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VirtualReality-pp
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Wrist Injury
Keywords: wrist injury; proprioception; virtual reality
MeSH Terms: conditions — Wrist Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional rehabilitation (Active Comparator): Conventional rehabilitation treatment for the wrist plus a specific proprioceptive exercise program.
  Interventions: Other: Rehabilitation treatment
- Rehabilitation+virtual reality (Experimental): Conventional rehabilitation treatment for the wrist plus a specific proprioceptive exercise program and virtual reality games
  Interventions: Other: Rehabilitation treatment; Other: Virtual Reality games

INTERVENTIONS:
Other: Rehabilitation treatment — ROM, strength, stretch and proprioception exercises
Other: Virtual Reality games — Virtual Reality games using META QUEST PRO glasses
  Arms: Rehabilitation+virtual reality

SUMMARY:
The goal of this randomized clinical trial is to compare how the incorporation of Virtual Reality could influence in proprioception, kinesiophobia, functionality and catastrophism in people that are undergoing a rehabilitation treatment after a wrist fracture. The principal questions it aims to answer are:

* Evaluate the effect of using virtual reality added to standard rehabilitation of wrist injuries in proprioception impairment.
* Evaluate the effect of using virtual reality on psychological factors as kinesiophobia and catastrofism.
* Evaluate the effect of using virtual reality in functionality on wrist-injured patients.

Intervention will be:

* Control group: participants of this group will receive conventional rehabilitation of the wrist, plus a specific proprioceptive exercise program.
* Experimental group: participants of this group will receive the same treatment as the control group but adding virtual reality games at the end of the session.

Researchers will compare control and experimental group to see if an implantation of Virtual Reality could had benefits on function, kinesiophobia, catastrofism and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Adult (equal or more than 18 y/o).
* Suffering wrist injury
* Agree and sign informed consent.

Exclusion Criteria:

* Not had suffered a wrist injury
* Suffer from any mental, cognitive, neurological or musculoskeletal disorder
* Have cervical pathology/impairment
* Have visual or balance problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proprioception | Baseline, 1 and 3 months
  Assessment of proprioception impairment using Joint Position Sense Test (JPST). Punctuation will be the difference between the asked position and the patient's replication. The test will be repeated with open and closed eyes.

SECONDARY OUTCOMES:
Kinesiophobia | Baseline, 1 and 3 months
  Fear of movement, assessed with Tampa Scale for Kinesiophobia (TSK) which has 17 items with Likert's answers. Punctuation goes from 17 to 68 points, where <37 points means a low level of kinesiophobia and >37 a high level.
Catastrophism | Baseline, 1 and 3 months
  Catastrophizing pain assessed with Pain Catasthrophizing Scale (PCS) which has 13 items with Likert's answers. Punctuation goes from 0 to 52 points, where 0-20 points means a low catastrophism, 21-30 points moderate catastrophism and >30 points a high catastrophism.
Function | Baseline, 1 and 3 months
  Functionality of the upper limb assessed with QuickDASH which has 11 items. Punctuation goes from 0 to 100, where 0 means no disability and 100 maximum disability.
Hand and Wrist function | Baseline, 1 and 3 months
  Assessed with Patient-Rated Wrist Evaluation (PRWE) which has 15 items punctuated from 0 to 10. Punctuation goes from 0-100 where 0 means no disability and 100 maximum disability.
Range of motion | Baseline, 1 and 3 months
  Range of motion of the wrist and fingers using a goniometer.
Force Sense | Baseline, 1 and 3 months
  GRIP's force sense assessed with Force Sense Test (FST), where punctuation is the difference between the asked and replicated force.